CLINICAL TRIAL: NCT03102736
Title: Pharmacologic Attenuation of Ketamine Using Nitroprusside
Brief Title: Ketamine and Nitroprusside for Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, MD, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 16-1580
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Depression
Keywords: depression; ketamine; nitroprusside
MeSH Terms: conditions — Depression | interventions — Ketamine; Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and research staff (aside from pharmacy) will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo and Ketamine (Placebo Comparator): Placebo saline given over 240 minutes + 0.5 mg/kg ketamine given over 40 minutes
  Interventions: Drug: Placebos; Drug: Ketamine
- Nitroprusside and Ketamine (Experimental): 0.5 mcg/kg/min nitroprusside given over 240 min (4 hours) - 0.5 mg/kg ketamine given over the last 40 min of the nitroprusside infusion (starting at minute 200 the two drugs are given together)
  Interventions: Drug: Ketamine; Drug: Nitroprusside

INTERVENTIONS:
Drug: Placebos — Placebo saline
  Arms: Placebo and Ketamine
Drug: Ketamine — 0.5 mg/kg ketamine
Drug: Nitroprusside — 0.5 mcg/kg nitroprusside
  Arms: Nitroprusside and Ketamine

SUMMARY:
The purpose of this study is to test the effects of the medication ketamine and the medication called nitroprusside in patients with major depression. Ketamine has both good and bad effects. Some studies have shown that ketamine improves depression. However, studies have also shown that it causes strange and sometimes unpleasant sensations referred to "psychotic" or "dissociative" symptoms. An example of a psychotic symptom would be hearing or seeing something that in reality is not there. The study team would like to see if nitroprusside can prevent the reported bad effects of ketamine without blocking the reported good effects. This might make ketamine a better treatment for depression.

DETAILED DESCRIPTION:
Ketamine is an effective fast-acting therapeutic intervention for patients with treatment refractory depression that is known to have the unwanted effect of inducing temporary psychotomimetic symptoms (i.e., delusions, hallucinations and thought disorganization) in some patients. The precise mechanisms of these psychotropic effects remain to be elucidated, but for several decades the NMDA-type glutamate receptor has been hypothesized to be of central importance. In this vain, recent studies of the antihypertensive agent nitroprusside - which increases the availability of the molecular nitric oxide, a known by-product of NMDA activity - have found evidence for antipsychotic properties both in humans with psychotic illness and healthy subjects given ketamine. Here, the clinical team proposes a study that will build on this work by evaluate the effects of nitroprusside on both the antidepressant and psychotomimetic effects of ketamine given to patients to treat refractory depression. In addition, as an exploratory aim, by collecting serial blood samples from the subjects, as the subjects are administered ketamine and nitroprusside, the clinical team will seek to determine functional markers of therapeutic effect and the mechanisms by which ketamine modulates both mood and psychotic states Research Question: The clinical team will test whether the effects of ketamine (KET) on mood and psychotic states is modified by co-administration with sodium nitroprusside (NP) in patients with depression. Furthermore, the clinical team will evaluate the extent to which the underlying biology of disease states and drug mechanisms can be inferred through analysis of brain-derived molecular material isolated from the peripheral circulation.

Specific Aims:

Aim I. To test whether co-administration with NP has any impact on the efficacy of KET as an antidepressant.

Aim II: To test the ability of NP to prevent the psychotomimetic effects of KET in patients with depression.

Research Hypotheses:

Research Hypothesis I. Patients pre-treated with NP will experience attenuated antidepressant effects (measured by MADRS score) following KET compared to pre-treatment with placebo.

Research Hypothesis II: Patients pre-treated with NP will experience attenuated psychotomimetic effects (e.g., CADSS score) immediately following KET compared to pre-treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 21-65 years of age;
* Female individuals who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or using a medically accepted reliable means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative pregnancy test at screening and at pre-infusion;
* Participants must fulfill current DSM-5 criteria for Major Depression without psychotic features or Persistent Depressive Disorder with specifier of "with persistent major depressive episode";
* Depression is at least moderate severity, defined as a CGI-S score of ≥ 4;
* Current major depressive episode is of at least 4 weeks duration
* Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document
* Each participant must be able to identify a family member, physician, or friend who will act as an emergency contact

Exclusion Criteria:

* Lifetime history of psychotic features, diagnosis of schizophrenia or any other psychotic disorder, or diagnosis of bipolar disorder;
* Lifetime histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
* Current diagnosis of obsessive compulsive disorder (OCD) or eating disorder (bulimia nervosa or anorexia nervosa);
* Subjects with DSM-V drug or alcohol abuse/dependence within the preceding 2 years;
* Patients with schizotypal or antisocial personality disorder, or any clinically significant axis II disorder that would, in the investigator's judgment, preclude safe study participation;
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk;
* Women who are either pregnant or nursing;
* Any serious, unstable medical illnesses including hepatic, renal impairment, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease;
* History of congestive heart failure or established coronary artery disease;
* History of cerebrovascular insufficiency
* History of intrapulmonary arteriovenous shunts, co-arctation of the aorta or other conditions where cardiac outflow tract is obstructed;
* Vitamin B12 deficiency;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Renal impairment, as reflected by a BUN > 20 mg/dL and/or creatinin clearance of >1.3 mg/dL;
* Thyroid impairment, as reflected by a thyroid-stimulating hormone (TSH) > 4.2 mU/L;
* Hepatic injury, as reflected by AST or ALT greater than twice the upper limit of the reference range (AST: >80; ALT >110)
* Patients who have a positive urine toxicology for illicit substances at screening and within 24 hours of the infusion;
* Treatment with an irreversible MAOI within 2 weeks prior to randomization or fluoxetine within 4 weeks prior to randomization;
* Treatment with other antidepressants (classified as SSRIs, SNRIs, Atypical Antidepressants, MAOIs, TCAs) within one week of randomization.
* Previous recreational use of phencyclidine (PCP) or KET;
* Hypertension with systolic BP >160 mm Hg or diastolic BP >90 mm Hg at screening, systolic BP > 165 mm Hg or diastolic BP > 95 mm Hg immediately prior to treatment with study drug or hypotension with systolic BP < 90 or diastolic < 60 at screening or immediately prior to treatment with study drug; heart rate >110 or <60 at either of these time points;
* Treatment with sildenafil (Viagra), tadalafil (Cialis), Avanafil (Stendra), Vardenafil (Levitra) or other drugs in the same category of phosphodiesterase-5 enzyme inhibitors within 2 weeks of infusion.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bevilacqua L, Charney A, Pierce CR, Richards SM, Jha MK, Glasgow A, Brallier J, Kirkwood K, Bagiella E, Charney DS, Murrough JW. Role of nitric oxide signaling in the antidepressant mechanism of action of ketamine: A randomized controlled trial. J Psychopharmacol. 2021 Feb;35(2):124-127. doi: 10.1177/0269881120985147. PMID 33522376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 participants enrolled, 14 were excluded before starting the study and 10 were excluded after starting the study but before randomization (6 were ketamine non-responder, 2, failed to return to baseline, and 2 withdrew before randomization)
Groups:
- Placebo and Ketamine: Placebo saline given over 240 minutes + 0.5 mg/kg ketamine given over the last 40 minutes of the infusion
Period: Overall Study
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (3.1) | 42.9 (11.7) | 37.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
MADRS [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Asberg Depression Rating Scale - This is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 (normal) and 60 (severe depression).
  units on a scale | 31.4 (5.3) | 26.9 (4.4) | 28.9 (5.2)
QIDS [Mean (Standard Deviation); unit: units on a scale] — Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) score - Each item is rated 0 (no depression) to 3 (severe depression). The total score ranges from 0-27, with higher score indicating more symptoms.
  units on a scale | 17.6 (3.6) | 14.3 (2.5) | 15.8 (3.4)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Full scale from 1-7, with higher score indication more symptoms.
  units on a scale | 4.7 (0.8) | 4.4 (0.5) | 4.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: This is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 (normal) and 60 (severe depression).
Time Frame: 24 hours after start of infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
Number analyzed (Participants) | 7 | 9
score on a scale | 13.4 (11.9) | 14.2 (10.2)

2. Secondary Outcome: Clinician-Administered Dissociative States Scale
Description: This is used to measure dissociative effects during the infusions. The scale includes 23 clinician administered items scored from 0 (not at all) to 4 (extremely). The CADSS measures impairment in body perception, environmental perception, time perception, memory impairment, and feelings of unreality. Full scale from 0-92, with lower score indicating better health outcomes.
Time Frame: 240 minutes after start of infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
Number analyzed (Participants) | 7 | 9
score on a scale | 11.5 (9.9) | 8.4 (4.1)

3. Secondary Outcome: Visual Analog Scale
Description: These scales are scored in millimeters from the left-hand side of a 100-mm line to a perpendicular mark made by the patient at a point corresponding to the apparent magnitude of the feeling state. Range: 0 ("not at all") to 100 ("most ever").
Time Frame: 240 minutes after start of infusion
Population: data not collected
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: BPRS used to assess acute behavioral changes during the infusions. Four key BPRS items for the positive (+) symptoms of psychosis will be used: conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content. Three items representing the negative (-) symptoms of psychosis will also be used: blunted affect, emotional withdrawal, and motor retardation. Each item scored 1-7. Full scale from 7 - 49, with higher score indicating more symptoms.
Time Frame: +240 minutes (after start of Placebo/Nitroprusside infusion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
Number analyzed (Participants) | 7 | 9
score on a scale | 7.5 (1.13) | 7.2 (0.66)

ADVERSE EVENTS:
Time Frame: 24 hours after infusion
Arm/Group | Placebo and Ketamine | Nitroprusside and Ketamine
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and Ketamine (N=7) | Nitroprusside and Ketamine (N=9)
Nausea (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Akathisia (Nervous system disorders) | 0 | 1
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Worsening MDD (Psychiatric disorders) | 0 | 1 — Major Depressive Disorder
Hypertension (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03102736/Prot_SAP_000.pdf